CLINICAL TRIAL: NCT04021992
Title: GVD±R (Gemcitabine, Oral Vinorelbine and Doxorubicin Liposome, With or Without Rituximab) Regimen for Autologous Hematopoietic Stem Cell Transplantation(ASCT)-Eligible Patients With Refractory/Relapsed Diffuse Large B-cell Lymphoma:a Multi-center, Single Arm, Phase II Study
Brief Title: GVD±R Regimen for ASCT-eligible Patients With Refractory/Relapsed DLBCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-088
Record Dates: First submitted 2019-07-13; First posted 2019-07-16 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Gemcitabine; Vinorelbine; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GVD with or without R (Experimental): Gemcitabine 1000mg/m2, d1,d8, intravenous drip; Vinorelbine 50mg/m2, d1,d8, oral; Doxorubicin liposomes 30mg/m2, d1,intravenous drip; With or without rituximab 375 mg/m2, d0,intravenous drip; All patients received up to 6 treatment cycles of 21 days.
  Interventions: Drug: gemcitabine, vinorelbine and doxorubicin liposome, with or without rituximab

INTERVENTIONS:
Drug: gemcitabine, vinorelbine and doxorubicin liposome, with or without rituximab — All patients enrolled in the study will accept gemcitabine, oral vinorelbine and doxorubicin liposome, with or without rituximab as their salvage chemotherapy.

SUMMARY:
The purpose of this multi-center,single arm,phase Ⅱ clinical trail is to determine the safety and efficacy of GVD±R (gemcitabine, oral vinorelbine and doxorubicin liposome, with or without rituximab) regimen for autologous hematopoietic stem cell transplantation(ASCT)-eligible patients with refractory/relapsed diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved CD20+ DLBCL;
* previously received at least one systemic treatment (including chemotherapy) without remission or relapse after remission;
* at least one evaluable lesion；
* ECOG PS 0-1;
* 18-65 years;
* proper functioning of the major organs.

Exclusion Criteria:

* involvement of central nervous system;
* with other malignancy;
* patients receiving or received drug of other clinical trial within 30 days；
* previously received doxorubicin liposome or have used other anthracycline drug with accumulated restricted doses (adriamycin 450mg/m2, epirubicin 935mg/m2, acrarubicin 900mg/m2)；
* patients who received treatment for hematologic toxicity caused by previous chemotherapy within 7 days before enrollment;
* grade 2 or more peripheral neuropathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
ORR | 4-years

SECONDARY OUTCOMES:
success rates in autologous stem cell mobilization | 4-years
PFS | 4-years
EFS | 4-years
OS | 4-years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China